CLINICAL TRIAL: NCT05370508
Title: A Phase 1/2 Dose Escalation and Expansion Study of Sonodynamic Therapy With SONALA-001 in Combination With Exablate 4000 Type 2.0 MR-Guided Focused Ultrasound in Subjects With Progressive or Recurrent Glioblastoma Multiforme (rGBM)
Brief Title: A Study of Sonodynamic Therapy Using SONALA-001 and Exablate 4000 Type 2.0 in Subjects With Recurrent GBM
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is terminated due to funding challenges and not due to safety concerns.
Sponsor: SonALAsense, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SDT-202; R44CA275508 (NIH)
Record Dates: First submitted 2022-05-04; First posted 2022-05-11 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Recurrent GBM
Keywords: Sonodynamic Therapy; SONALA-001; Exablate 4000 Type 2.0; MR-guided Focused Ultrasound; SDT; rGBM; Aminolevulinic acid HCI; ALA HCI; ALA
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (5):
- Cohort 1 (Experimental): 10 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 1
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 2 (Experimental): 10 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 2
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 3 (Experimental): 10 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 3
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 4 (Experimental): 10 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 4
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 5 (Experimental): Recommended Phase 2 Dose (RP2D) IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 5
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)

INTERVENTIONS:
Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS) — SONALA-001(ALA) given 6-12 hours prior to receiving the MRgFUS
  Other Names: Exablate Type 2.0

SUMMARY:
The primary objectives of this trial are to evaluate the safety, dose-limiting toxicities, maximum tolerated dose (MTD), maximum administered dose (MAD) and recommended Phase 2 dose (RP2D) for future study after a single treatment of SONALA-001 in combination with MRgFUS and to evaluate preliminary efficacy of sonodynamic therapy (SDT) using SONALA-001 and Exablate Type 2.0 device in subjects with progressive or recurrent GBM.

ELIGIBILITY:
Inclusion Criteria

1. Must be 18 years or older at the screening visit.
2. Histologically proven GBM (as defined in 2021 WHO Classification of Tumors of the Central Nervous System; Louis, Perry, et al. 2021) that has recurred or progressed, and for which resection is not indicated.
3. Tumor must be located in the supratentorial or cerebellar region. Tumors with infratentorial locations require consultation with the Sponsor/Medical Monitor to confirm suitability for treatment.
4. Previous treatment with standard of care radiotherapy (RT) and temozolomide (temozolomide required only if tumor has at least partial methylation of the O6-methylguanine-DNA methyltransferase promoter). Temozolomide should be administered concurrent with RT and adjuvantly for newly diagnosed disease unless intolerant or ineligible for treatment.
5. No recurrence within 4 weeks of completion of RT, defined from the imaging assessment immediately after completion of RT.
6. Up to two prior systemic treatments for recurrent or progressing disease.
7. If receiving corticosteroids, must be maintained on a stable or decreasing dosage of steroids for at least 7 days prior to C1D1.
8. Karnofsky Performance Score (KPS) ≥ 70 assessed within 14 days of C1D1.
9. Must have adequate organ and marrow function as defined below:

   * Absolute neutrophil count ≥ 1.5 ×10⁹/L (1,500/μL), without the use of myeloid growth factors (e.g., granulocyte-colony stimulating factor) within 7 days prior to C1D1 for short acting growth factors and 14 days for long-acting growth factors to meet eligibility.
   * Platelets ≥ 75 × 10⁹/L (100,000/μL), unsupported, defined as no platelet transfusion within 7 days prior to C1D1.
   * Hemoglobin ≥ 9 g/dL maintained without the need for erythropoietin stimulating agents; subjects that require transfusion or growth factors need to demonstrate stable hemoglobin of ≥ 9 g/dL over at least a 7-day period immediately prior to C1D1.
   * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN), in subjects with Gilbert syndrome, total bilirubin >1.5 ULN as long as direct bilirubin is normal.
   * ALT (SGPT) < 3 x institutional ULN.
   * AST (SGOT) < 3 x institutional ULN.
   * Albumin ≥ 3 g/dl.
   * Potassium ≥ lower limit of normal (LLN).
   * Serum total calcium (correct for serum albumin) or ionized calcium ≥ LLN.
   * Estimated creatinine clearance (CrCl) by the Cockcroft-Gault (C-G) equation or measured ≥ 60 mL/min. Actual body weight will be used for calculation of the C-G equation. If estimated CrCl is abnormal, accurate measurement should be obtained by 24-hour urine collection to measure CrCl.
10. All colony-forming growth factor(s) (i.e., filgrastim, sargramostim or erythropoietin) must have been discontinued for at least 7 days prior to C1D1 or 14 days if pegylated (PEG) formulations were received.
11. Have a life expectancy of at least 12 weeks.
12. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
13. Ability to provide written, signed, and dated (personally or via a legally authorized representative) informed consent at screening as applicable to participate in the study.
14. Females of childbearing potential (FOCP) must have a negative serum pregnancy test at screening. Subjects of childbearing or child-fathering potential must be willing to use highly effective birth control during the entire study. Acceptable forms of birth control include hormonal contraceptives (oral, depot, injectable, transdermal, or intravaginal) or intrauterine device (IUD) for at least one week prior to study treatment, condom and spermicidal or diaphragm and spermicidal. Other acceptable forms of birth control include a) abstinence for subjects who are not sexually active or b) if the subject is in a monogamous relationship with a partner who is sterile (e.g., vasectomy performed at least 6 months prior to subject's first study treatment). Subjects who become sexually active or begin to have relations with a partner who is not sterile during the trial must agree to use an effective form of birth control for the duration of the study. FOCP taking hormonal therapy must be on treatment for at least 12 weeks prior to C1D1 and must not change their dosing regimen during the study.

Exclusion Criteria

Target disease

1. Tumor in the brainstem (not including fluid-attenuated inversion recover [FLAIR] changes), or a diagnosis of gliomatosis cerebri (highly infiltrative T2 hyperintense tumor with ill-defined margins encompassing at least three lobes of the brain). Tumors with infratentorial locations require consultation with the Sponsor/Medical Monitor to confirm suitability for treatment.

   Concurrent or prior therapy
2. Subjects who have not recovered to Grade 1 or baseline from AEs (CTCAE v 5.0, or most current) related to prior anticancer therapy (excluding alopecia, lymphopenia, peripheral neuropathy, and ototoxicity, which are excluded only if ≥ Grade 3).
3. Prior systemic anticancer treatment:

   1. Chemotherapy, biologic therapy (i.e., small molecular inhibitors), monoclonal antibodies, investigational agents) within 21 days or 5 half-lives (whichever is shorter), prior to C1D1 or per below:
   2. Nitrosoureas or bevacizumab within 2 weeks prior to C1D1
   3. If a subject is receiving an anti-PD-1 or anti-PD-L1 antibody on a shorter frequency (i.e., every two weeks), then the subject is eligible if last dose was within 2 weeks prior to C1D1.
4. Prior therapy such as interstitial brachytherapy, Gliadel® Wafers (carmustine implants), laser interstitial thermal therapy (LITT), or Optune therapy, within 4 weeks prior to C1D1 or as long as there are any ongoing treatment-related CTCAE Grade ≥2 AEs or intolerable side effects.
5. Radiation therapy within 4 weeks prior to C1D1.
6. Use of potentially phototoxic substances (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, tetracyclines, sulfonamides, quinolones, hypericin extracts, topical preparations containing ALA) within 24 hours before and after SONALA-001 infusion.
7. Use of fish oil supplements within 24 hours of C1D1 is allowed if the subject's clotting parameters fall within normal limits.
8. Use of blood thinning agents within 7 days prior to C1D1. Subjects whose medical condition does not permit discontinuation of this therapy are excluded.
9. Prior major surgery within 3 weeks prior to C1D1. Major surgery is defined as any significantly invasive procedure into a major body cavity (abdomen, cranium etc.) and/or surgery requiring extensive recuperation (joint replacement). Please discuss with the Sponsor/Medical Monitor if there are any questions.

   Medical history and concurrent disease
10. Diagnosis of porphyria.
11. Hypersensitivity to porphyrins.
12. Known history of allergy to gadolinium contrast agents.
13. Inability to undergo MRI (e.g., verify the model of the pacemaker for ability to be used with MRI).
14. Malignant disease, other than that being treated in this study. Note: Subjects with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g., breast carcinoma, cervical cancer in situ) that have undergone potentially curative therapy are not excluded. Other exceptions include malignancies that were treated curatively and have not recurred within 2 years prior to C1D1 and any malignancy considered indolent or that do not require therapy.
15. Significant acute deterioration in neurologic status within 7 days prior to C1D1, in the opinion of the investigator, including but not limited to new onset seizures and/or increasing doses of corticosteroids.
16. Uncontrolled concurrent illness including, but not limited to:

    * ongoing or active infection.
    * transfusion dependent thrombocytopenia or anemia that prevent meeting hematological inclusion criteria.
    * psychiatric illness/social situations that would limit compliance with study requirements.
17. Clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormality.
18. Pregnancy or breastfeeding.
19. A known or underlying medical condition that, in the opinion of the investigator or Sponsor, could make the administration of investigational drug/ study treatment hazardous to the subject, or could adversely affect the ability of the subject to comply with or tolerate the study.
20. Inability to participate in the opinion of the investigator, by being unwilling or unable to return for required follow-up visits or to obtain follow-up studies to assess toxicity to therapy or to adhere to study plan, procedures, and restrictions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-07-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability of SONALA-001 SDT as assessed by the frequency and severity of dose-limiting toxicities (DLTs) | Day 1 to Day 21 post treatment
  Safety and tolerability of SONALA-001 SDT
  Definitions of Dose Limiting Toxicities (DLTs):
  The DLT window is the 21-day period following the first study treatment per patient.
  DLTs are defined as the following events during the DLT window, not clearly related to underlying disease, disease progression or intercurrent illness, as determined by safety review committee:
  Any death
  Non-hematologic toxicity:
  Any CTCAE Grade 3 or higher Hy's law cases Moderate heating/burning at the scalp Grade 3 or greater neurological toxicities Evidence of clinically significant tissue damage outside the region targeted by MRgFUS Grade 3 or greater photosensitivity in subjects strictly following restrictions to light exposure to sunlight or room lights for 48 hours after SONALA-001 administration
  Hematologic toxicity:
  Grade 4 neutropenia for more than 7 days Grade 3 or higher thrombocytopenia with clinically significant bleeding Neutropenic fever
Safety and Tolerability of SONALA-001 SDT as assessed by the number of subjects with Adverse Events (AEs), adverse device effects (ADEs), serious AEs (SAEs) and serious device effects (SADEs) | Day 1 to 12 months
  Safety and tolerability of SONALA-001 SDT
  Definition of Adverse Event (AE) An AE is defined as the appearance of (or worsening of any pre-existing) undesirable sign(s), symptom(s), or medical condition(s) that occur after the first dose of investigational drug. Abnormal laboratory values or test results occurring after the first dose of investigational drug constitute AEs only if they induce clinical signs or symptoms, are considered clinically significant, require therapy (e.g., hematologic abnormality that requires transfusion or hematological stem cell support) except electrolytes which require replacement therapy and correct to CTCAE grade ≤ 1 within 48 hours unless considered life-threatening, or require changes in study medication(s).
Safety and Tolerability of SONALA-001 SDT as assessed by the number of subjects with abnormal hematology, chemistry, coagulation and urinalysis laboratory tests. | Day 1 to 12 months
  Lab tests covered by CTCAE version 5.0 or most current will be graded accordingly. For lab tests covered by CTCAE, a Grade 0 will be assigned for all non-missing values not graded as 1 or higher. Grade 5 will not be used. For lab tests where grades are not defined by CTCAE, results will be categorized by low/normal/high classifications based on lab normal ranges or categorized by normal/abnormal for character (descriptive) lab values.
To determine Maximum Administered Dose (MAD), Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) after a single treatment of MR-guided Focused Ultrasound (MRgFUS) energy in combination with SONALA-001 SDT (Phase 1) | Up to 3 weeks post treatment
  Determination of Recommended Phase 2 Dose of SONALA-001 SDT in combination with MRgFUS
Progression-free survival rate at 6 Months (Phase 2) | 6 Months
  To evaluate preliminary efficacy (PFS rate at 6 months) of the RP2D of ALA SDT treatments by mRANO in subjects with recurrent GBM
Safety of the RP2D of ALA SDT as assessed by the number of subjects with AEs/ADEs, SAEs/SADEs, abnormal laboratory tests, neurologic and physical examinations, vital signs, and ECGs. | Day 1 to 12 months
  Safety of the RP2D of ALA SDT

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating Area Under the plasma Concentration (AUC) vs. time from time 0 to the last measurable time point (AUC-t) (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating AUC for plasma concentration vs. time from time 0 to infinity (AUC0-∞) (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating AUC for plasma concentration vs. time from time 0 to time to maximum drug concentration (Tmax) (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating AUC for plasma concentration vs. time from time 0 to time to terminal elimination half-life (t½) (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating AUC for plasma concentration vs. time from time 0 to time to clearance. (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001 by calculating AUC for plasma concentration vs. time from time 0 to time to elimination rate constant. (Phase 1) | Day 1 to 24 hours post SONALA-001 dosing
  Samples will be collected at 12 time points during 24 hours pre/post SONALA-001 administration.
To evaluate the preliminary antitumor activity Objective Response Rate (ORR): Complete Response (CR) and Partial Response (PR) by mRANO | Day 1 to 12 months
  ORR defined as the proportion of subjects with a best overall response (BOR) of CR or PR as assessed per mRANO by investigator assessment
To evaluate preliminary efficacy and Duration of Response (DOR) (Phase 1) | Up to 12 months
  DOR, defined as time from date of first documented objective response (CR or PR) to the first documented progression or death due to any cause.
To evaluate preliminary efficacy and Overall Survival (OS) (Phase 1) | Up to 12 months
  OS, defined as time from first dose of study treatment to death due to any cause.
To evaluate preliminary efficacy and clinical benefit rate Clinical Benefit Rate (CBR) (Complete Response (CR), Partial Response (PR), and Stable Disease (SD) | Up to 12 months
  CBR defined as the proportion of subjects with a BOR of CR or PR or SD.
To evaluate preliminary efficacy and Duration of Clinical Benefit (DOCB) (Phase 2) | Up to 12 months
  DOCB defined as time from date of first documented objective response (CR or PR) and SD to first documented progression or death due to any cause.
To evaluate preliminary efficacy and Time To Response (TTR) | Up to 12 months
  TTR, calculated as time from first dose of study treatment to first documented objective response (CR or PR).
To evaluate preliminary efficacy and Progression Free Survival (PFS) | Up to 12 months
  PFS defined as time from first dose of study treatment to progression or death due to any cause.
To evaluate preliminary efficacy and PFS rate at 6 and 12 months | Up to 12 months
  PFS rate at 6 months (Phase 1) and 12 months defined as the percentage of subjects without progression or death at 6 months and 12 months.
To evaluate preliminary efficacy and and OS (Phase 2) | Up to 12 months
  OS, defined as time from first dose of study treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Andresen, MD, Study Director — SonALAsense, Inc.
Locations (6):
- United States (6):
  - Ivy Brain Tumor Center, Phoenix, Arizona
  - UCSF, San Francisco, California
  - Mayo Clinic, Rochester, Minnesota
  - NYU Langone Health, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No